CLINICAL TRIAL: NCT04065009
Title: A Randomized Double Blind, Multicenter Trial to Assess Time-interval Between Cytoreductive Surgery and Adjuvant Chemotherapy After Administration of Local Anesthetic Intraperitoneally/Perioperatively in Advanced Epithelial Ovarian Cancer
Brief Title: The IPLA-OVCA Trial, Intra-Peritoneal Local Anaesthetics in Ovarian Cancer
Acronym: IPLA-OVCA
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Skane University Hospital (Other)
Responsible Party: Principal Investigator, Sahar Salehi, Senior Consultant, Assistant Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 20190729
Record Dates: First submitted 2019-08-19; First posted 2019-08-22 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Advanced Ovarian Cancer
Keywords: Local Anesthesia; Time-interval from surgery to adjuvant chemotherapy; advanced ovarian cancer
MeSH Terms: interventions — Ropivacaine; Saline Solution

STUDY DESIGN:
Intervention Model Description: Randomised, double blind, prospective, multicenter
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study drugs are blinded and administered perioperatively. Fully blinded for all (participants, assessors etc)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Normal saline administered intraperitoneally at defined times during upfront surgery and intermittently postoperatively for 72 hours
  Interventions: Drug: Saline Solution
- Experimental (Experimental): Local anesthetic (ropivacaine) administered intraperitoneally at defined times during upfront surgery and intermittently postoperatively for 72 hours
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine — Experimental drug will be administered intraperitoneally
  Other Names: Narop
  Arms: Experimental
Drug: Saline Solution — Placebo will be administered intraperitoneally
  Other Names: Normal saline
  Arms: Placebo

SUMMARY:
Surgery and chemotherapy combined constitute first line treatment in women with advanced ovarian cancer. The aim of surgery apart from staging is cytoreduction, i.e. surgical resection of tumour. Radical resection of all tumour visible by the naked eye followed by adjuvant chemotherapy is associated with best chance of prolonged survival. However, because of tumour dissemination in the peritoneal cavity, radical surgery is often very extensive with surgery in all quadrants of the abdomen and multi-organ resection with substantial risk of postoperative severe complications and subsequent delay in administration of adjuvant chemotherapy. Longer time-interval between surgery to start of adjuvant chemotherapy has been associated with decrease in survival.

Surgery presents opportunities not only for eradicating tumours but, paradoxically, also for proliferation and invasion of residual cancer cells. It increases the shedding of malignant cells into the blood and lymphatic circulations, inhibits their apoptosis and potentiates their invasion capacity. Additionally, the immune system, the inflammatory system and the neuroendocrine system react to surgery with important changes, which have been proven to promote progression of cancer. Several anaesthesia-related factors play an important role in perioperative tumorigenesis such as inhalational anaesthetics, opiate analgesics, local anaesthetics and regional anaesthesia, all of which may impact short-term morbidity and long-term mortality. A previous randomized placebo-controlled pilot study suggests that women who receive local anesthetics intraperitoneally preoperatively have a significantly decreased time-interval to initiation of adjuvant chemotherapy.

In a prospective, randomised, multi-centre study, we plan to further assess if intraperitoneal local anaesthetics administered perioperatively during 72 h leads to early start of chemotherapy compared to placebo in patients undergoing cytoreductive surgery for FIGO stage III-IV ovarian cancer.

DETAILED DESCRIPTION:
Epithelial ovarian cancer (EOC) is the common term for cancer that originate from the surface of the ovary, lining of the fallopian tube and the peritoneum. There are different histopathological subtypes with high grade serous adenocarcinomas being the most prevalent (70%) followed by endometrioid (10%), clear cell (10%), low-grade serous (5%) and mucinous adenocarcinomas (3%).The pattern of dissemination is foremost through early exfoliation or seeding of tumour-cells in the peritoneum (carcinomatosis) and the majority of women have advanced stage disease at presentation, why ovarian cancer is the gynecologic malignancy with highest mortality.

Ovarian cancer affects 295 000 women every year globally and causes 185 000 cancer-related deaths annually . The highest incidence is seen in Northern Europe and North America and the lowest in South East Asia and parts of Africa. In the Nordic countries 2300 women are diagnosed annually and the corresponding number in Sweden is 700. Ovarian cancer constitutes 3% of all female cancers in Sweden and the risk of developing disease before the age of 75 is 1.1%. A decline in incidence is evident since the 1970s most probably due to increase in use of contraceptive pills but also change in criteria for diagnosis (an adnexal biopsy is mandatory for diagnosis today). The median age at diagnosis is 63 years.

Risk-factors include genetic mutations, family history, hormone replacement therapy and endometriosis. Pregnancy, lactation, contraceptive pills, sterilization, salpingectomy, hysterectomy and salpingoophorectomy are all factors associated with decreased risk of developing EOC.

Staging of ovarian cancer is surgical and according to the International Federation of Gynecology and Obstetrics (FIGO), latest revised in 2014 (7). In stage III and IV, advanced ovarian cancer, extra-pelvic dissemination is evident. Stage of disease is a strong prognostic factor for survival. The total 5-year relative survival in Sweden is 50% but ranges from 90% for stage I to 20% for stage IV. However, treatment is also an important prognostic factor and may increase survival even in advanced stage.

Surgical treatment of advanced EOC is often accompanied by a severe inflammatory and immuno-compromised perioperative course associated with early morbidity, delayed rehabilitation and, sometimes, delayed start of chemotherapy. Early start of chemotherapy has been repeatedly associated with improved survival. For this reason, perioperative factors such as choice of anaesthesia and analgesia and fluid replacement may be important.

Tumorigenesis and the perioperative environment Surgery, perioperative stress and anaesthesia may all modulate the immuno-surveillance mechanisms and compromise host defences that normally maintain a balance between immunity & tumorigenesis. There is increasing evidence that surgery itself may promote the recurrence and metastases of cancer, which depends largely on the tumour's ability to metastasise, combined with the host immunity and inflammatory response. Natural killer (NK) cells act as a primary defence against perioperative cancer metastases. Negative effects of anaesthetics and analgesics on NK-cell activity may promote pro-inflammatory effects and may also activate cancer cell survival pathways. Additionally, concentrations of tumour-related anti-angiogenic factors are decreased while angiogenic factors such as vascular endothelial growth factor (VEGF) are increased. Hypoxia inducing factor (HIF-1) is a transcriptional factor that has also been shown to play an important role for tumour survival. Hypoxia in solid tumours leads to activation of HIF-1, which in turn increases cancer cell survival . Similarly, hyperoxia may, paradoxically, lead to activation of HIF-1 and potentially worsen long-term survival. Inhalational anaesthetics but not propofol have been shown to affect VEGF as well as transforming growth factor-beta (TGF-β) in patients undergoing breast surgery that may affect long-term survival. VEGF and TGF-β play a significant role in establishing tumour blood supply and cell proliferation. Other factors such as surgical stress, blood transfusions, hypothermia, hyperglycaemia, and postoperative pain may also affect immunity and the tumour microenvironment.

Role of anaesthetics and analgesics in cancer metastases Preventing a major systemic inflammatory response and preserving immuno-surveillance in the perioperative period are fundamental in promoting improved postoperative outcome in cancer surgery. The severity of injury correlates with the magnitude of inflammation. In vitro studies have shown that amide local anaesthetics have cytotoxic activity, which could prove to be beneficial in preventing cancer recurrence. These potential cytotoxic effects of LA may effectively reduce postoperative morbidity and promote early start of chemotherapy. Anaesthetic drugs, specifically inhalation anaesthetics, impair numerous immune functions, including those of neutrophils, macrophages, dendritic cells, T-cell, and natural killer (NK) cells. Upregulation of hypoxia-inducible-factors (HIF) in tumour cells by volatile anaesthetics may contribute to a tumour's recurrence by stimulating cytoprotective or pro-tumorigenic behaviour in residual cells. However, propofol may not depress the immune function and does not upregulate synthesis of HIF. Opioid analgesics inhibit both cellular and humoral immune function, increase angiogenesis, and promote breast tumour growth in rodents. Opioids interfere with immune function by depressing NK cell activity . The use of epidural anaesthesia and analgesia thus prevents the stress response to surgery, reduces the need for opiates and may prolong survival.

Fluid dynamics and early recovery Fluid optimization remains a challenge because of several factors: preoperative fluid shifts and accumulation of ascitic fluid, low preoperative albumin from malnutrition, as well as perioperative fluid and blood loss. Both hypo- and hypervolemia have been shown to have adverse effects and may delay recovery and start of chemotherapy and a large prospective, randomised study concluded that hypovolemia may even lead to renal insufficiency.

The primary objective of this Phase 3 double blind placebo controlled trial is to investigate if local anesthetics administered intraperitoneally perioperatively at time of upfront surgery for advanced ovarian cancer reduces the time-interval between surgery and adjuvant chemotherapy.

Secondary objectives are to investigate, postoperative morbidity, complications and long term survival.

The trial entails a translational part with the following specific aims:

I. To examine if surgical peritoneal stress evolves during the course of surgery, as measured by pro-inflammatory cytokines and biomarkers in the mesothelium, tumour tissues and blood, coupled to analysis of the circulating tumour DNA II. To test if intraperitoneally administered anti-inflammatory analgesics may reduce the (mesothelial) inflammation.

III. To use functional ex vivo assays for exploring how the above identified surgical tissue responses and induced or inhibited pathways affect the aggressive EOC cell functions and properties including tumour invasion and chemo-resistance.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III
* Scheduled for upfront cytoreductive surgery for presumed stage III or IV epithelial ovarian cancer
* Signed written informed consent

Exclusion Criteria:

* Contraindication to epidural anesthesia
* Allergy to any component drugs used during epidural or intraperitoneal anesthesia (Ropivacaine, Sufentanil)
* Uncontrolled renal, liver, heart failure or ischemic heart disease
* Speech, language or cognitive difficulties
* Women in whom cytoreductive surgery is not attempted at time of upfront laparotomy due to extent of disease

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2020-08-26 (Actual); Primary Completion 2024-01-10 (Estimated); Study Completion 2028-08-26 (Estimated)

PRIMARY OUTCOMES:
Time-interval from upfront surgery to adjuvant chemotherapy | Number of days to start of adjuvant chemotherapy (0 - 60 days)
  Days from surgery to first infusion of adjuvant chemotherapy

SECONDARY OUTCOMES:
Postoperative complications | 30 days postoperatively
  Assessed according to the Clavien-Dindo Nomenclature
Overall survival | 3 and 5 years after surgery
  Death of any reason
Postoperative quality of recovery | Perioperatively
  As measured by validated instruments
Postoperative morbidity | Perioperatively
  As measured by validated instruments

CONTACTS AND LOCATIONS:
Overall Officials: Sahar Salehi, MD, PhD, Principal Investigator — Karolinska Institute and Karolinska University Hospital
Locations (1):
- Karolinska Hospital, Solna, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
All study data will be retained at site of patient recruitment. Primary investigator and statistician will only have access to coded patient identity

REFERENCES:
- [Background] Hayden JM, Oras J, Block L, Thorn SE, Palmqvist C, Salehi S, Nordstrom JL, Gupta A. Intraperitoneal ropivacaine reduces time interval to initiation of chemotherapy after surgery for advanced ovarian cancer: randomised controlled double-blind pilot study. Br J Anaesth. 2020 May;124(5):562-570. doi: 10.1016/j.bja.2020.01.026. Epub 2020 Mar 13. PMID 32172954
- [Derived] Hasselgren E, Kofoed NG, Falconer H, Bjorne H, Zach D, Hunde D, Johansson H, Asp M, Thorlacius K, Kannisto P, Salehi S. Prospective Assessment of Clinically Relevant Fluid Balance Thresholds Associated With Postoperative Complications in Advanced Ovarian Cancer. Acta Anaesthesiol Scand. 2025 Oct;69(9):e70112. doi: 10.1111/aas.70112. PMID 40856042
- [Derived] Gultekin O, Gonzalez-Molina J, Sarhan D, Groes-Kofoed N, Hassan MU, Lehti K, Salehi S. Systemic and tumor-specific inflammatory markers VCAM-1 and ICAM-1 as indicators of extent of surgery and oncologic outcome in advanced ovarian cancer. Transl Oncol. 2025 Sep;59:102462. doi: 10.1016/j.tranon.2025.102462. Epub 2025 Jul 12. PMID 40652770
- [Derived] Hasselgren E, Groes-Kofoed N, Falconer H, Bjorne H, Zach D, Hunde D, Johansson H, Asp M, Kannisto P, Gupta A, Salehi S. Effect of intraperitoneal ropivacaine during and after cytoreductive surgery on time-interval to adjuvant chemotherapy in advanced ovarian cancer: a randomised, double-blind phase III trial. Br J Anaesth. 2025 Mar;134(3):662-670. doi: 10.1016/j.bja.2024.10.015. Epub 2024 Nov 20. PMID 39572271